CLINICAL TRIAL: NCT04386473
Title: Comparison of Cardiac Function Between Left Bundle Branch Pacing and Right Ventricular Outflow Tract Septal Pacing in Pacemaker-dependent Patients
Status: Completed | Type: Observational
Sponsor: Ruiqin xie (Other)
Responsible Party: Sponsor-Investigator, Ruiqin xie, director of cardiology department, The Second Hospital of Hebei Medical University
Organization: The Second Hospital of Hebei Medical University (Other)
Other Study IDs: XieruiqindoctorLBBP
Record Dates: First submitted 2020-05-06; First posted 2020-05-13 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2020-05

CONDITIONS: Slow Arrhythmia; Left Bundle Branch Pacing; Cardiac Function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Left Bundle Branch Pacing
  Interventions: Device: pacemaker
- Right Ventricular Outflow Tract Septal Pacing
  Interventions: Device: pacemaker

INTERVENTIONS:
Device: pacemaker — electrode is implanted in left bundle branch in LBBP; electrode is implanted in right ventricular outflow tract septal in RVOP

SUMMARY:
Permanent pacemaker implantation is a common method for bradycardia and cardiac conduction dysfunction. With the development of physiological pacing, the optimal location of ventricular pacing site is still improving. Traditional ventricular pacing site at the apex of right ventricle or septum of right ventricular outflow tract（RVOT）, causing iatrogenic left bundle branch block and asynchronous ventricular contraction, leading to cardiac remodeling, pacemaker-mediated cardiomyopathy and congestive cardiac failure. Long-term chronic ventricular pacing can lead to changes in endocardial myocytes and myofibrils and promote fibrosis. Thus, the alternative pacing site, HIS bundle pacing, has been sought later. The safety and feasibility of permanent HIS bundle pacing have been confirmed in patients with various cardiac diseases. However, the shortcomings of high and unstable threshold, long implantation time, low R-wave amplitude and HIS bundle damage during implantation limit the application of HIS pacing especially in patients with infra-Hisian block. Left bundle branch pacing(LBBP) is a new technique evolved from HIS bundle pacing. In 2017, Huang et al[9]reported that LBBP was successfully paced using 3830 leads(Medronic Inc. USA). The advantages of narrow QRS duration, low threshold, high R wave amplitude, easy fixation and correction of left bundle branch block made LBBP more widely used in clinic.However, whether left bundle branch pacing is superior to traditional right ventricular outflow tract septal pacing in cardial function is still lack of sufficient evidence. The purpose of this study is aim to using Brain natriuretic peptide(BNP), echocardiography and speckle-tracking echocardiagraphy, six minutes walk test and quality of life to compare the changes of cardiac function within 1 month between LBBP and RVOP in pacemaker-dependent patients.

DETAILED DESCRIPTION:
The purpose of this study was to compare the changes of cardiac function within 1month in pacemaker-dependent patients between LBBP and RVOP. A single-center prospective random controlled clinical study was conducted in 60 patients with bradycardia indications. 30 patients underwent RVOP and 30 patients underwent LBBP. The changes of BNP, echocardiogram and speckle-tracking echocardiagraphy, six minutes walk test and quality of life were compared between the two groups before and within 1month. The etiology of pacemaker implantation included high atrioventricular block, atrial fibrillation with slow arrhythmia. Implantation procedures: Left bundle branch pacing was achieved by trans-interventricular septum method in the basal ventricular septum and performed by using the Select pacing 3830 lead(Medtronic Inc, USA) delivered through a fixed sheath(7F C315 HIS, Medtronic Inc, USA). During implantation, a unipolar configuration is used for pacing and recording. The delivery sheath was inserted through left subclavian vein into atrial side of the tricuspid valve to mark His bundle potential under right anterior oblique(20°) fluoroscopic view. As a marker in His bundle region, the sheath with the lead tip was further advanced towards the right side of the ventricular septum approximately 1.5-2cm, and paced QRS morphology showing left bundle branch block(LBBB) at output of 2V/0.4ms. When the sheath with the lead tip screwed to the left side of the septum, paced QRS morphology changed from LBBB to right bundle branch block(RBBB), a gradual change of the notch morphology("W" waveform) in lead V1 gradually shifted and finally disappeared.Another active electrode is implanted in the right auricle.Patients with RVOP: The right ventricular pacing lead was positioned in the low intervals of right ventricular outflow tract, and atrial active lead was positioned at right auricle. BNP was measured routinely before implantation and reexamined on 1 day and 1month after pacemaker implantation.Twelve-lead ECG were recorded including QRS duration, QRS amplitude and QT interval. Echocardiography data were measured by conventional transthoracic echocardiography system including left atrial anteroposterior dimension, left atrial transverse dimension, left atrial vertical dimension, e', peak E-wave velocity, peak A-wave velocity, E/A, E/e', left atrial ejection fraction (LAEF), left ventricular ejection fraction (LVEF), velocity-time integration of aortic blood flow(VTI). Left atrial strain and strain rate were measured by speckle-tracking echocardiography(STE).We also measure the six minutes walk test and quality of life in all patients before and after implantation in 1month.

ELIGIBILITY:
Inclusion Criteria:

Pacemaker-dependent patients who agreed to implant a pacemaker.

Exclusion Criteria:

Patients with congenital heart diseases, such as atrial septal defect, ventricular septal defect, or rheumatic heart diseases, valvular heart diseases.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pacemaker-dependent patients who agreed to implant a pacemaker.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Changes in B natriuretic peptide | baseline, 1 day and 1month after implantation
  Blood samples are extracted in all patients to detected
Changes in Electrocardiograph | baseline, 1 day and 1 month after implantation
  QRS duration in ms, QT duration in ms
Changes of the Data of Pacemaker | baseline and 1month after implantation
  Threshold value in V, sense in mV of the pacemaker
Changes of Ultrasonic Cardiogram | baseline, 7 days and 1 month after implantation
  UCG:sizes of LA in mm
Changes of Ultrasonic Cardiogram | baseline, 7 days and 1 month after implantation
  ejection fraction of LV and LA (%)
Changes of six minutes walk test | baseline, 7 days and 1 month after implantation
  six minutes walk test in meter.
Changes of quality of life | baseline and 1 month after implantation
  SF-36 quality of life test.

CONTACTS AND LOCATIONS:
Locations (1):
- Second Hospital of Hebei Medical University, Shijiazhuang, Hebei, China